CLINICAL TRIAL: NCT03522584
Title: Durvalumab (MEDI4736), Tremelimumab and Palliative Hypofractionated Image Guided Radiation Therapy (HIGRT) in Patients With Recurrent/Metastatic Squamous Cell Carcinomas of the Head and Neck Previously Treated With Immune Checkpoint Inhibitors
Brief Title: Durvalumab, Tremelimumab and Hypofractionated Radiation Therapy in Treating Patients With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated by the sponsor due to lack of efficacy in study treatment.
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Cristina Rodriguez, Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9881; NCI-2018-00540 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9881 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG1717067 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Results first posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Metastatic Head and Neck Squamous Cell Carcinoma; Recurrent Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — durvalumab; Immunoglobulin G; Disulfides; Radiosurgery; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Treatment (tremelimumab, durvalumab, HIGRT, SBRT) (Experimental): Patients receive tremelimumab IV over 1 hour and durvalumab IV over 1 hour on day 1, week 1. Treatment repeats every 4 weeks for up to 4 cycles or every 6 weeks for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive durvalumab IV over 60 minutes on day 1, week 16. Treatment repeats every 4 weeks for up to 9 cycles or every 6 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo hypofractionated radiation therapy using either HIGRT or SBRT over 3 fractions QOD during week 3.
  Interventions: Biological: Durvalumab; Other: Laboratory Biomarker Analysis; Radiation: Stereotactic Body Radiation Therapy; Biological: Tremelimumab; Procedure: Hypofractionated Image-Guided Radiation Therapy

INTERVENTIONS:
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
Other: Laboratory Biomarker Analysis — Correlative studies
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy
Biological: Tremelimumab — Given IV
  Other Names: Anti-CTLA4 Human Monoclonal Antibody CP-675,206; CP-675; CP-675,206; CP-675206; Ticilimumab
Procedure: Hypofractionated Image-Guided Radiation Therapy — Undergo HIGRT
  Other Names: Hypofractionated Image-Guided Radiotherapy

SUMMARY:
This phase I/II trial studies the side effects of durvalumab, tremelimumab and hypofractionated radiation therapy in treating patients with head and neck squamous cell carcinoma that has come back (recurrent) or that has spread to other places in the body (metastatic). Immunotherapy with monoclonal antibodies, such as durvalumab and tremelimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Hypofractionated radiation therapy delivers higher doses of radiation therapy over a shorter period of time and may kill more tumor cells and have fewer side effects. Giving durvalumab, tremelimumab, and hypofractionated radiation therapy may work better in treating patients with recurrent or metastatic head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To demonstrate safety and tolerability of durvalumab and tremelimumab and palliative radiation therapy in patients with recurrent metastatic squamous cell carcinomas of the head and neck previously exposed to an anti PD-1 or PDL-1 monoclonal antibody.

SECONDARY OBJECTIVES:

I. Measure objective response rates based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. criteria in patients receiving the durvalumab, tremelimumab and palliative radiation therapy (RT) combination.

II. Determine overall and progression free survival in patients enrolled in the study.

OUTLINE:

Patients receive tremelimumab intravenously (IV) over 1 hour and durvalumab IV over 1 hour on day 1, week 1. Treatment repeats every 4 weeks for up to 4 cycles or every 6 weeks for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive durvalumab IV over 60 minutes on day 1, week 16. Treatment repeats every 4 weeks for up to 9 cycles or every 6 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo hypofractionated radiation therapy using either hypofractionated, image-guided radiotherapy (HIGRT) or stereotactic body radiation therapy (SBRT) over 3 fractions every other day (QOD) during week 3.

After completion of study treatment, patients are followed up at 30 days, 2, 3, 4, 6, 8, and 10 months, and then every 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven recurrent/metastatic squamous cell carcinoma arising from a previous head and neck primary site, and located within the head and neck region, lung mediastinum, lymph nodes, soft tissue metastases or bone, and who are not candidates for curative intent therapy
* An actual body weight > 40kg
* Demonstrated disease progression during, or after discontinuation, of the most recent line of systemic therapy
* Have received any number lines of prior systemic therapy (including systemic therapy in the curative intent setting, and including a platinum containing regimen)
* Have received an anti-PD1 or anti PDL1 monoclonal antibody
* Have a target lesion/s deemed suitable by the treating physicians for hypofractionated radiation therapy (HIGRT or SBRT) with the intent of palliation or prevention of symptoms; this lesion must be: a) 1-3 non overlapping sites in the head and neck region OR b) metastatic lesions outside the head and neck (H&N) region in the lung mediastinum, soft tissue metastases, lymph nodes or bone (a minimum of 1 and a maximum 5 lesions will be irradiated), provided there is no significant overlap between the lesions; patients should have RECIST 1.1 criteria measurable disease in addition to the lesion/s treated with radiation; if the site/s of radiation were previously radiated to high dose RT (> 50 Gy), there should be > 6 month time interval between the last dose of radiation and the start of radiation
* Have the ability to tolerate required radiotherapy-related procedures (e.g.: lie flat and hold position for treatment) as determined by the treating physician
* Be willing and able to provide written informed consent for the trial and comply with the study visit requirements
* Have measurable disease based on RECIST 1.1. (in addition to the lesion/s that will be treated with hypofractionated radiation therapy)
* Have provided tissue from an archival tissue sample or newly obtained core or excisional biopsy of a tumor lesion
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Hemoglobin >= 9.0 g/dL (should be performed within 10 days of treatment initiation)
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (>= 1500 per mm^3) (should be performed within 10 days of treatment initiation)
* Platelet count >= 100 x 10^9/L (>= 100,000 per mm^3) (should be performed within 10 days of treatment initiation)
* Serum bilirubin =< 1.5 x institutional upper limit of normal (ULN) (should be performed within 10 days of treatment initiation); this will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be =< 5 x ULN (should be performed within 10 days of treatment initiation)
* Serum creatinine clearance (CL) > 60 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance (should be performed within 10 days of treatment initiation)
* Evidence of post-menopausal status OR negative urinary or serum pregnancy test for female pre-menopausal patients; women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause; the following age-specific requirements apply:

  * Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy, or hysterectomy)
  * Women >= 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
* Female subjects of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 1 method of highly effective birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 180 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 180 days after the last dose of study therapy
* Patient is >= 5 years free of another primary malignancy, except: a) if the other malignancy is basal cell carcinoma or cervical carcinoma in situ or b) if the other primary malignancy is not considered clinically significant and is requiring no active intervention

Exclusion Criteria:

* Has a body weight =< 40kg at the time of enrollment
* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment
* Has a target lesion/s for radiotherapy that is > 5 cm (> 50 cc) in greatest dimension
* Has a target lesion/s in a region that previously received high dose radiation therapy (RT) (> 50 Gy) demonstrating any of the following:

  * carotid artery encasement (> 180 degrees)
  * unprotected carotid artery (i.e. skin is directly over the carotid without intervening soft tissue, especially after prior neck dissection without a vascularized free flap) (a&b due to risk of carotid blow out)
  * skin infiltration by tumor (due to risk of fistula)
  * located in the larynx/hypopharynx primaries (due airway threat)
  * treated with high dose radiation therapy (> 50 Gy) within 6 months or less of trial enrollment
* Any prior grade >= 3 immune-related adverse event (irAE) while receiving a prior immunotherapy agent, or any unresolved irAE > grade 1
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab; the following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., computed tomography [CT] scan premedication)
* Has received a prior monoclonal antibody within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has received prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: Subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Has known brain metastases or spinal cord compression unless the patient is stable (asymptomatic; no evidence of new or emerging brain metastases; and stable and off steroids for at least 14 days prior to start of study treatment); following radiotherapy and/or surgery of the brain metastases patients must wait 4 weeks following the intervention and before initiating study treatment with imaging to confirm stability
* Has an active autoimmune disease requiring systemic treatment within the past 2 years or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents; subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule; subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study; subjects with hypothyroidism stable on hormone replacement will not be excluded from the study
* Has evidence of current interstitial lung disease (ILD) or pneumonitis or a prior history of ILD or pneumonitis requiring oral or intravenous glucocorticoids
* Has an active infection requiring systemic therapy
* Requires therapeutic anticoagulation or has known active bleeding diathesis
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 180 days after the last dose of trial treatment
* Has received prior therapy with an anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has evidence of acute or chronic hepatitis B or hepatitis C
* Has received a live vaccine within 30 days prior to the first dose of trial treatment
* Has a mean QT interval corrected for heart rate (QTc) >= 470ms calculated from 3 electrocardiograms (ECGs) using Fridericia's Correction
* Has a history of primary immunodeficiency or an allogeneic organ transplant
* Has a history of hypersensitivity to durvalumab or tremelimumab excipient
* Known history of previous clinical diagnosis of tuberculosis
* Uncontrolled intercurrent illness including, but not limited to symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2022-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristina P. Rodriguez, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Tremelimumab, Durvalumab, HIGRT, SBRT)
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Tremelimumab, Durvalumab, HIGRT, SBRT)
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 64 [47 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Effects Graded According to Common Terminology Criteria for Adverse Events (CTCAE) v. 4.0
Description: Toxicities will be summarized as the number and percentage of patients with each type of toxicity, per Criteria for Adverse Events version 4.0
Time Frame: From the start of study treatment up to 3 months after last study treatment, up to 38 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Tremelimumab, Durvalumab, HIGRT, SBRT)
Number analyzed (Participants) | 6
Participants
  Anorexia | 1
  Concentration Impairment | 1
  Cough | 2
  Depression | 1
  Diarrhea | 1
  Dizziness | 1
  Dry Mouth | 1
  Fatigue | 4
  Fever | 2
  Headache | 2
  Hypercalcemia | 1
  Hyperalbuminemia | 1
  Increased Dyspnea | 1
  Non-Cardiac Chest Pain | 1
  Infusion Related Reaction | 1
  Mucositis | 1
  Nausea | 1
  Neck Pain | 1
  Night Sweats | 1
  Otitis Externa | 1
  Pruritus | 1
  Right Shoulder Pain | 1
  Maculopapular Rash | 1
  Rhinorrhea | 1
  Shingles | 1
  Sore Throat | 1
  Weight Loss | 3
  Wheezing | 1
  Oral Thrush | 1

2. Secondary Outcome: Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Tremelimumab, Durvalumab, HIGRT, SBRT)
Number analyzed (Participants) | 5
Participants
  Stable Disease | 3
  Progressive Disease | 1
  Complete Response | 1

3. Secondary Outcome: Progression-free Survival
Description: Survival estimates will be calculated using the Kaplan-Meier method. Progression free survival is measured in months. PFS is defined as the amount of time between treatment initiation and when the disease progresses per RECIST 1.1 criteria
Time Frame: From the date of study enrollment for up to 2 years
Measure: Median (Standard Deviation); unit: months
Arm/Group | Treatment (Tremelimumab, Durvalumab, HIGRT, SBRT)
Number analyzed (Participants) | 6
months | 7 (2)

4. Secondary Outcome: Overall Survival
Description: Survival estimates will be calculated using the Kaplan-Meier method. Overall survival is measured in months. OS is defined as the amount of time between treatment initiation and when the patient is deceased.
Time Frame: From the date of study enrollment for up to 2 years
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Tremelimumab, Durvalumab, HIGRT, SBRT)
Number analyzed (Participants) | 6
months | 8 [4 to 14]

ADVERSE EVENTS:
Time Frame: 3 years, 2 months
Description: Adverse events and serious adverse events will be recorded from time of administration of the first dose of investigational drug, throughout the treatment period and including the follow-up period (90 days after the last dose of durvalumab + tremelimumab).
Arm/Group | Treatment (Tremelimumab, Durvalumab, HIGRT, SBRT)
All-Cause Mortality (participants affected / at risk) | 6/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Tremelimumab, Durvalumab, HIGRT, SBRT) (N=6)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Concentration Impairment (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Depression (Nervous system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1)
Dry Mouth (Metabolism and nutrition disorders) | 1 (1)
Fever (Infections and infestations) | 2 (2)
Headache (General disorders) | 2 (2)
Hypercalcemia (Endocrine disorders) | 1 (1)
Hyperalbuminemia (Endocrine disorders) | 1 (1)
Increased Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Non-Cardiac Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Night Sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Otitis Externa (Musculoskeletal and connective tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2)
Right Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Maculopapular Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Shingles (Infections and infestations) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Weight Loss (Metabolism and nutrition disorders) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oral Thrush (Infections and infestations) | 1 (1)
Fatigue (General disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-10): https://cdn.clinicaltrials.gov/large-docs/84/NCT03522584/Prot_SAP_001.pdf